CLINICAL TRIAL: NCT06926374
Title: Prospective Evaluation of Cornerstone Robotics Sentire Surgical System in Major Gastrointestinal and Urologic Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Simon S. M. Ng, Wei Lun Professor of Surgery, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CREC 2025.109-T
Record Dates: First submitted 2025-04-07; First posted 2025-04-13 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Colorectal Carcinoma; Rectal Prolapse; Prostate Cancer (Adenocarcinoma); Bladder Cancer; Kidney Cancer; Hiatal Hernia With Gastroesophageal Reflux Disease; GIST - Gastrointestinal Stromal Tumor; Esophageal Cancer; Gallstones; Gastric Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Prolapse; Prostatic Neoplasms; Adenocarcinoma; Urinary Bladder Neoplasms; Kidney Neoplasms; Gastrointestinal Stromal Tumors; Esophageal Neoplasms; Gallstones; Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Robotic surgery using the Sentire Surgical System (Experimental): Robotic surgery using the Sentire Surgical System
  Interventions: Procedure: Robotic surgery using the Sentire Surgical System

INTERVENTIONS:
Procedure: Robotic surgery using the Sentire Surgical System — Robotic surgery using the Sentire Surgical System

SUMMARY:
Robotic assisted surgery has been performed for more than two decades with good success and safety profile. However, there was only one dominating robotic surgical system available in the past which led to high cost for robotic surgery. Recently, a new robotic surgical system (Sentire Robotic Surgical System) was introduced by researchers of The Chinese University of Hong Kong (CUHK). This new robotic surgical system aims to achieve similar outcomes and standards of robotic surgery performed using the dominating system but with a significantly lower cost. The technologic innovation and development of this new robotic system is made by the Cornerstone Robotics Limited, which is based in Hong Kong. In a pilot clinical study conducted at Prince of Wales Hospital involving 55 patients, the Sentire Robotic Surgical System had demonstrated high success rate with minimal complications in patients who underwent robotic colorectal, upper gastrointestinal, and urologic surgery. Researchers of CUHK would therefore like to conduct another prospective study to further evaluate the efficacy and safety of Sentire Surgical System C1000 in major gastrointestinal and urologic surgery with expanded indications. It is believed that the results of this study will provide data to support its use for wide range of procedures with minimal access trauma, for the benefit of patients. This system will also lead to a wider range of clinical application for minimally invasive surgery with a cost-effective model.

DETAILED DESCRIPTION:
As above.

ELIGIBILITY:
General Inclusion Criteria for All Procedures:

* Body mass index <35 kg/m2
* Suitable for the listed minimally invasive surgical procedures for treatment of respective diseases
* Willingness to participate as demonstrated by giving informed consent

General Exclusion Criteria for All Procedures:

* Contraindication to general anesthesia
* Severe concomitant illness that drastically shortens life expectancy or increases risk of therapeutic intervention
* Untreated active infection
* Noncorrectable coagulopathy
* Presence of another malignancy or distant metastasis
* Emergency surgery
* Vulnerable population (e.g., mentally disabled, pregnancy)

Robotic Colorectal Resection

Inclusion Criteria:

- Adenocarcinoma or large adenoma (not amenable to endoscopic removal) located at the colorectum (from the cecum to the anal verge) amenable to minimally invasive surgery

Exclusion Criteria:

* T4 tumor
* Recurrent tumor
* Extensive previous abdominal surgery precluding minimally invasive surgery

Robotic Transanal Total Mesorectal Excision

Inclusion Criteria:

- Mid/low rectal adenocarcinoma located <12 cm from the anal verge

Exclusion Criteria:

* T4 tumor or involvement of circumferential resection margin even after neoadjuvant therapy
* Tumor requiring multivisceral resection
* Tumor requiring abdominoperineal resection; recurrent rectal tumor
* T1 tumor that can be treated by local excision
* Extensive previous abdominal surgery

Robotic Rectopexy

Inclusion Criteria:

* Clinically diagnosed with previously untreated and uncomplicated rectal prolapse or enterocele

Exclusion Criteria:

- Extensive previous abdominal surgery precluding minimally invasive surgery

Radical Prostatectomy

Inclusion Criteria:

- Clinically diagnosed with nonmetastatic adenocarcinoma of prostate

Exclusion Criteria:

- Previous history of prostate surgery (e.g., transurethral resection of prostate)

Total or Partial Nephrectomy

Inclusion Criteria:

- Clinically diagnosed with nonmetastatic kidney cancer

Exclusion Criteria:

* Previous ipsilateral kidney surgery
* Complex kidney anatomy (e.g., horseshoe kidney, complex renal vascular anatomy)

Radical Cystectomy

Inclusion Criteria:

- Clinically diagnosed with nonmetastatic bladder cancer

Robotic Esophageal Hiatal Surgery and Fundoplication

Inclusion Criteria:

- Clinically diagnosed with Hiatal Hernia and / or Gastroesophageal reflux disease amendable to fundoplication

Exclusion Criteria:

- Previous history of laparotomy precluding minimally invasive surgery

Robotic Gastrectomy

Inclusion Criteria:

- Clinical diagnosis of gastric tumor (Adenocarcinoma or Gastrointestinal Stromal Tumor (GIST)) amendable to minimally invasive radical gastrectomy

Exclusion Criteria:

- Previous history of laparotomy precluding minimally invasive surgery

Robotic Esophagectomy

Inclusion Criteria:

- Clinical diagnosis of carcinoma of esophagus amendable to minimally invasive esophagectomy

Exclusion Criteria:

- Esophageal carcinoma after definitive chemoradiotherapy and indicated for salvage esophagectomy

Robotic Cholecystectomy

Inclusion Criteria:

- Symptomatic gallbladder stones clinically indicated for laparoscopic cholecystectomy

Exclusion Criteria:

* Acute cholecystitis
* Previous history of abdominal surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Conversion rate | Up to 1 month
  The definition of a conversion for this study is an emergent change in the treatment plan to conventional minimally invasive (laparoscopic/thoracoscopic) surgery (i.e., the use of more than one additional port), multiport robotic surgery, or to open surgery.
Perioperative complications | Up to 1 month
  Perioperative complications including intraoperative complications and all complications occurring during the hospital stay or within 30 days after discharge will be graded according to the Clavien-Dindo classification. Complications of Clavien-Dindo grade III (those requiring surgical, endoscopic, or radiologic intervention) or above are regarded as major complications.

SECONDARY OUTCOMES:
Operative time | Up to 1 month
Operative blood loss | Up to 1 month
Pain scores on a visual analog scale | Up to 1 month
Analgesic requirement | Up to 1 month
Length of hospital stay | Up to 1 month
Resection margin positivity for malignancy | Up to 1 month
Number of lymph nodes harvested | Up to 1 month
Anal continence after surgery, measured by the Cleveland Clinic Incontinence Score (Wexner's Score) | Up to 12 months
  The Cleveland Clinic Incontinence Score or Wexner's Score is the most common score used to determine the severity of incontinence before and after surgery for anal incontinence. The scoring system takes into account the type and frequency of incontinence, and the extent to which it alters the patient's life. It consists of five questions to assess the degree of incontinence (solid, liquid, gas, wears pad, lifestyle alteration). The frequency of each type of incontinence is rated on a scale ranging from 0 (never) to 4 (always or to once a day) so that the sum of the frequencies add up to a total score that may range from 0 to 20. Higher scores indicate higher levels of incontinence.
Male sexual function after surgery, measured by the International Index of Erectile Dysfunction - 5 (IIEF-5 questionnaire) | Up to 12 months
  IIEF-5 is an abridged five-item version of the 15-item International Index of Erectile Function (IIEF) which is used to diagnose the presence and severity of erectile dysfunction. This questionnaire consists of only five questions and each IIEF-5 item is scored on a five-point ordinal scale where lower values represent poorer sexual function. Thus, a response of 0 for a question is considered the least functional, whereas a response of 5 is considered the most functional. The possible scores for the IIEF-5 range from 1 to 25 (one question has scores of 1-5), and a score above 21 is considered as normal erectile function and at or below this cutoff, erectile dysfunction.
Urinary function after surgery, measured by the International Prostate Symptom Score (IPSS) | Up to 12 months
  IPSS is based on the answers to seven questions concerning urinary symptoms and one question concerning quality of life. Each question concerning urinary symptoms allows the patient to choose one out of six answers indicating increasing severity of the particular symptom. The answers are assigned points from 0 to 5. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic).

CONTACTS AND LOCATIONS:
Overall Officials: Simon SM Ng, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, The Chinese University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No